CLINICAL TRIAL: NCT02360527
Title: Retinal Neurodegeneration in Type 2 Diabetes as Biomarker for Alzheimer´s Disease
Acronym: DIALRET
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(IR)15/2014
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Retinal Neurodegeneration; Alzheimer´s Disease; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Biochemical evaluation including Hba1c, lipidic profile, renal and hepatic function. We will also determine the APOE genotype and plasmatic beta-amyloidal fractions (Aβ1-40 and Aβ1-42) as previously described (Hixson JE and Vernier DT. Restriction isotyping of human apolipoprotein E by gene amplification and cleavage with HhaI. J Lipid Res 1990;31:545-8.)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Type 2 diabetic patients with AD: 35 patients
- Type 2 diabetic patients with MCI: 35 patients
- Type 2 diabetic patients controls: 35 patients
- Non-diabetic patients with AD: 35 patients

SUMMARY:
A clear association between type 2 diabetes (T2D) and Alzheimer's disease (AD) has been reported. This association is independent of vascular impairment, and therefore, it could be attributed to neurodegeneration triggered or accelerated by diabetes itself. At present there are no methods to identify T2D patients at risk for developing AD. The retina shares many features with the brain and, therefore, has been suggested as an easily accessible way of examining pathology in the brain. In fact, many patients with AD present retinal abnormalities. However, the diagnosis of diabetes, a condition frequently associated with retinal neurodegeneration, has not been considered. On this basis, the final aim of this proposal is to identify diabetic patients at risk for developing AD based on the assessment of retinal neurodegeneration by means of non-invasive tests. Specific aims: 1) To compare the prevalence of morphological and functional abnormalities related to retinal neurodegeneration among three groups of T2D patients: patients with AD, patients with Mild Cognitive Impairment (MCI) and patients without AD or MCI. 2) To assess whether the retinal neurodegenerative features are related to severity of AD. 3) To explore whether the combined retinal neurodegeneration in diabetic patients with AD has a different functional and/or morphological pattern in comparison with neurodegeneration secondary to diabetes alone. Methods: Case-control study. Retinal neurodegeneration will be assessed by mutifocal electroretinogram (mfERG) and spectral domain optical coherence tomography (SD-OCT). The potential confounders will be considered in data analyses. Feasibility: A unique multidisciplinary consortium has been created in order to warrant the feasibility of the project Expected impact: This innovative approach will fill a gap that currently exist in the health care system and will reduce the economic burden associated with T2D patients with AD. In addition, this project would be the backbone for future prospective studies.

DETAILED DESCRIPTION:
A case control study in the recruitment will be carried out from the Diabetes outpatient clinic of a tertiary hospital (HUVH) and from the ACE Foundation. The investigators will include the following groups: 1) Type 2 diabetic patients with AD; B) Type 2 diabetic patients with MCI; 3) Type 2 diabetic patients with normal cognitive status; 4) Non-diabetic patients with AD. The groups will be matched by age (± 5 years), gender, risk factors related to AD (APOE genotype and family history of dementia), diabetes duration and Hba1c (±1%)- the last two criteria apply for the three groups of diabetic patients. Inclusion criteria: Written informed consent obtained from the patient; Age >65years; Diabetes duration>5 years; HbA1c < 10%; No apparent or mild non-proliferative DR according to the International Clinical Diabetic Retinopathy Disease Severity Scale. Exclusion criteria: Patients with other neurodegenerative diseases of the brain or retina (i.e. glaucoma) or cerebrovascular diseases. Sample size calculation: Assuming that diabetic patients will present around 30% of abnormal mfERG implicit time, and considering that this figure will be up 60% in those diabetic patients with AD, the number of patients required in each group would be 25. This calculation has been performed taking into account a 2-side risk level of 0.05 and a statistical power of 80%. However, it should be noted that this estimation has been performed taken into account the variables concerning AD. Therefore, it is foreseeable that more patients will be needed to obtain valid results for MCI. Consequently, the investigators feel it reasonable to extend the sample to 35 subjects per group.

The study will be divided into two stages (as will be further detailed): -Stage I: This will be the first step of the project and type 2 diabetic patients with AD and patients with normal cognitive status will be compared. -Stage II: Type 2 diabetic patients with MCI will be compared with patients with normal cognitive status or AD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the patient; Age >65years; Diabetes duration>5 years; HbA1c < 10%; No apparent or mild non-proliferative DR according to the International Clinical Diabetic Retinopathy Disease Severity Scale

Exclusion Criteria:

* Patients with other neurodegenerative diseases of the brain or retina (i.e. glaucoma) or cerebrovascular diseases.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will include the following groups: 1) Type 2 diabetic patients with AD; B) Type 2 diabetic patients with MCI; 3) Type 2 diabetic patients with normal cognitive status; 4) Non-diabetic patients with AD. The groups will be matched by age (± 5 years), gender, risk factors related to AD (APOE genotype and family history of dementia), diabetes duration and Hba1c (±1%)- the last two criteria apply for the three groups of diabetic patients.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Retinal neurodegeneration among three groups of type 2 diabetic patients patients with AD, patients with MCI and patients without AD or MCI. | 9 month
  -To compare the prevalence of morphological (SD-OCT) and functional abnormalities (mfERG) related to retinal neurodegeneration among three groups of type 2 diabetic patients: patients with AD, patients with MCI and patients without AD or MCI. In addition, a group of non diabetic subjects with AD will also be included.
  These groups will be matched by age, gender, duration of diabetes, HbA1C, and genetic risk factors for AD.
  * To assess whether the retinal neurodegenerative features are related to the severity of AD.
  * To explore whether the combined retinal neurodegeneration in diabetic patients with AD has a different functional and/or morphological pattern in comparison with neurodegeneration secondary to diabetes alone.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Hernandez, MD, PhD, Principal Investigator — Vall d´Hebron Research Institute VHIR
Locations (1):
- Vall d´Hebron Research Institute VHIR, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ciudin A, Simo-Servat O, Hernandez C, Arcos G, Diego S, Sanabria A, Sotolongo O, Hernandez I, Boada M, Simo R. Retinal Microperimetry: A New Tool for Identifying Patients With Type 2 Diabetes at Risk for Developing Alzheimer Disease. Diabetes. 2017 Dec;66(12):3098-3104. doi: 10.2337/db17-0382. Epub 2017 Sep 26. PMID 28951388